CLINICAL TRIAL: NCT03455816
Title: Randomized Clinical Study to Evaluate the Bio-Psychosocial Impact of a Mobile App for Diabetes ("SOCIAL DIABETES") and a SMARTMETER® (A. MENARINI DIAGNOSTICS) in the Care of People With Diabetes Mellitus Type 1 and Its Associated Costs
Brief Title: Clinical Study to Evaluate the Bio-Psychosocial Impact of Mobile App for Diabetes Type 1 ("SOCIAL DIABETES")
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soledad Ruiz de Adana (Other)
Responsible Party: Sponsor-Investigator, Soledad Ruiz de Adana, Maria Soledad Ruiz de Adana, Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud
Organization: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Social Diabetes
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: mobile app
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group that uses the Social Diabetes App (research group) (Experimental): This group use the App Social diabetes with the glucometer Glucomen Areo to monitoring the glucemia during 6 month
  Interventions: Device: Social Diabetes App
- Usual clinical monitoring group (control group) (Active Comparator): This group does not use the App. This group have an intermediate visit at 3 months with de doctor to see blood glucose self-monitoring and propose adjustments
  Interventions: Device: Usual clinical monitoring group (Control group)

INTERVENTIONS:
Device: Social Diabetes App — Social diabetes is an app for diabetes, free with CE mark, that by means of the incorporation of a glucometer ("glucomen Areo") allows through NFC technology the automatic introduction of data in the application
  Arms: Group that uses the Social Diabetes App (research group)
Device: Usual clinical monitoring group (Control group) — Active Comparator: Usual clinical monitoring group (control group) This group does not use the App. This group have an intermediate visit at 3 months with de doctor to see blood glucose self-monitoring and propose adjustments
  Arms: Usual clinical monitoring group (control group)

SUMMARY:
Based on international recommendations, the current clinical research project considers the effectiveness of a free diabetes app with a CE (Conformité Européenne) mark, "Social Diabetes", which incorporates the addition of a glucometer ("Glucomen Areo") it allows using NFC technology the automatic introduction of data, evaluating the impact on metabolic results and other related psychosocial variables, in people with diabetes 1 through a randomized randomized study during 6 months of follow-up.

DETAILED DESCRIPTION:
Randomized study in people with type 1 diabetes in intensive insulin therapy MDI with analogues and with HbA1c> 7% to the usual clinical follow-up options (CG) vs use of Social Diabetes App (GI) for 6 months.

The current clinical research project considers the effectiveness of a free diabetes app with a CE mark, "Social Diabetes", which incorporates the addition of a glucometer ("Glucomen Areo") it allows using NFC (Near Field Communication) technology the automatic introduction of data, evaluating the impact on metabolic results and other related psychosocial variables, in people with diabetes 1.

The substitution of the usual face-to-face medical visit every 3-4 months by the incorporation of an app system has a similar effect in terms of glycemic control (measured through HbA1c) in patients with DM1 treated with multiple doses of insulin per day (MDI). ) and inadequate metabolic control (HbA1c> 7%). In addition, it could save costs and consumption of health resources, and improve both the quality of life and the satisfaction of people with DM1.

The present study will be carried out under the usual conditions of clinical practice.

No pharmacological intervention, other than the usual clinical practice, will be applied to the included patients.

The people with diabetes 1 included in the study have a profile of "expert patient" having completed their diabetological education program at basic and advanced level (count of rations, calculations of ratios and sensitivity indexes) in such a way that the application will only be an aid in your daily decision making (mathematical calculations of ratios, IS, and recommended insulin doses, which you usually have to do "by hand").

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM1 over 1 year evolution.
* Age ≥18 and <65 years.
* HbA1c prior to the inclusion of the study> 7%.
* Intensive insulin treatment with MDI in basal-bolus regimen.
* Patients with basic digital skills and with 3G mobile phone and NFC technology.
* Patients who have given their informed consent in writing.

Exclusion Criteria:

* Treatment with subcutaneous insulin infusor (ISCI)
* Chronic kidney disease, liver disease, thyroid dysfunction (except hypothyroidism correctly treated and controlled).
* Pregnancy or pregnancy planning.
* Diabetes mellitus type 2.
* Severe psychological alterations.
* Absence of collaboration (informed consent).
* Patients who are participating in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
glycosylated hemoglobin | 6 month
  Metabolic impact measured through HbA1c of a mobile application (Social Diabetes) in the care of people with DM1.
Quality of life assessment: Diabetes Quality of Life (DQoL) questionnaire. | 6 month
  34 items to analyze the biopsychosocial impact measured through the quality of life questionnaire (DQol) of a mobile application (Social Diabetes) in the care of people with DM1.

SECONDARY OUTCOMES:
Mean blood glucose | 6 month
  Glycemic control: Mean blood glucose measured in mg / dl
Standard deviation | 6 month
  Glycemic variability: Standard deviation ( SD)
Number of mild hypoglycaemia | 6 month
  Number of mild hypoglycemia in two weeks
Number of severe hypoglycaemia | 6 month
  Number of severe hypoglycaemia in the last 6 months
Number of hyperglycemia | 6 month
  Number of hyperglycemia greater than 250mg / dl in two weeks
Episodes of ketosis | 6 month
  Number of episodes of ketosis in the last 6 months
Episodes of ketoacidosis | 6 month
  Number of episodes of ketoacidosis in the last 6 months
Number of hospital admissions for glycemic decompensation | 6 month
  Number of hospital admissions for glycemic decompensation in the last 6 months.
Fear of hypoglycemia: Questionnaire FH-15 | 6 month
  Fear of hypoglycemia: measured with the FH-15 scale. 15 items related to the fear of hypoglycemia in patients with type 1 diabetes.
Diabetes treatment satisfaction questionnaire ( DTSQ) | 6 month
  8 items concerning the satisfaction of the treatment
Diabetes distress scale. DDS | 6 month
  17 items on the problems and stress that people with type 1 diabetes suffer (Polonski y col,2005)
Scale of adherence to treatment in patients with diabetes type 1 | 6 month
  15 items related to adherence to patient treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Regional University Hospital of Málaga, Málaga, Spain

REFERENCES:
- [Background] Lewis TL, Boissaud-Cooke MA, Aungst TD, Eysenbach G. Consensus on use of the term "App" versus "Application" for reporting of mHealth research. J Med Internet Res. 2014 Jul 17;16(7):e174; discussion e174. doi: 10.2196/jmir.3460. No abstract available. PMID 25033233
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Franc S, Daoudi A, Mounier S, Boucherie B, Dardari D, Laroye H, Neraud B, Requeda E, Canipel L, Charpentier G. Telemedicine and diabetes: achievements and prospects. Diabetes Metab. 2011 Dec;37(6):463-76. doi: 10.1016/j.diabet.2011.06.006. Epub 2011 Sep 1. PMID 21889388
- [Background] Stone AA, Shiffman S, Schwartz JE, Broderick JE, Hufford MR. Patient non-compliance with paper diaries. BMJ. 2002 May 18;324(7347):1193-4. doi: 10.1136/bmj.324.7347.1193. No abstract available. PMID 12016186
- [Background] Holtz B, Lauckner C. Diabetes management via mobile phones: a systematic review. Telemed J E Health. 2012 Apr;18(3):175-84. doi: 10.1089/tmj.2011.0119. Epub 2012 Feb 22. PMID 22356525
- [Background] Chomutare T, Fernandez-Luque L, Arsand E, Hartvigsen G. Features of mobile diabetes applications: review of the literature and analysis of current applications compared against evidence-based guidelines. J Med Internet Res. 2011 Sep 22;13(3):e65. doi: 10.2196/jmir.1874. PMID 21979293
- [Background] Charpentier G, Benhamou PY, Dardari D, Clergeot A, Franc S, Schaepelynck-Belicar P, Catargi B, Melki V, Chaillous L, Farret A, Bosson JL, Penfornis A; TeleDiab Study Group. The Diabeo software enabling individualized insulin dose adjustments combined with telemedicine support improves HbA1c in poorly controlled type 1 diabetic patients: a 6-month, randomized, open-label, parallel-group, multicenter trial (TeleDiab 1 Study). Diabetes Care. 2011 Mar;34(3):533-9. doi: 10.2337/dc10-1259. Epub 2011 Jan 25. PMID 21266648
- [Background] Kirwan M, Vandelanotte C, Fenning A, Duncan MJ. Diabetes self-management smartphone application for adults with type 1 diabetes: randomized controlled trial. J Med Internet Res. 2013 Nov 13;15(11):e235. doi: 10.2196/jmir.2588. PMID 24225149
- [Background] Vahatalo M. Cellular phone transferred self blood glucose monitoring: Prerequisites for positive outcome. Practical Diabetes International 2004;21(5):192-194.
- [Background] Gomez EJ, Hernando Perez ME, Vering T, Rigla Cros M, Bott O, Garcia-Saez G, Pretschner P, Brugues E, Schnell O, Patte C, Bergmann J, Dudde R, de Leiva A. The INCA system: a further step towards a telemedical artificial pancreas. IEEE Trans Inf Technol Biomed. 2008 Jul;12(4):470-9. doi: 10.1109/TITB.2007.902162. PMID 18632327
- [Background] Benhamou PY, Melki V, Boizel R, Perreal F, Quesada JL, Bessieres-Lacombe S, Bosson JL, Halimi S, Hanaire H. One-year efficacy and safety of Web-based follow-up using cellular phone in type 1 diabetic patients under insulin pump therapy: the PumpNet study. Diabetes Metab. 2007 Jun;33(3):220-6. doi: 10.1016/j.diabet.2007.01.002. Epub 2007 Mar 28. PMID 17395516
- [Background] Cafazzo JA, Casselman M, Hamming N, Katzman DK, Palmert MR. Design of an mHealth app for the self-management of adolescent type 1 diabetes: a pilot study. J Med Internet Res. 2012 May 8;14(3):e70. doi: 10.2196/jmir.2058. PMID 22564332
- [Background] Froisland DH, Arsand E, Skarderud F. Improving diabetes care for young people with type 1 diabetes through visual learning on mobile phones: mixed-methods study. J Med Internet Res. 2012 Aug 6;14(4):e111. doi: 10.2196/jmir.2155. PMID 22868871
- [Background] Piette JD. Interactive behavior change technology to support diabetes self-management: where do we stand? Diabetes Care. 2007 Oct;30(10):2425-32. doi: 10.2337/dc07-1046. Epub 2007 Jun 22. No abstract available. PMID 17586735
- [Background] Montori VM, Helgemoe PK, Guyatt GH, Dean DS, Leung TW, Smith SA, Kudva YC. Telecare for patients with type 1 diabetes and inadequate glycemic control: a randomized controlled trial and meta-analysis. Diabetes Care. 2004 May;27(5):1088-94. doi: 10.2337/diacare.27.5.1088. PMID 15111526
- [Background] Liang X, Wang Q, Yang X, Cao J, Chen J, Mo X, Huang J, Wang L, Gu D. Effect of mobile phone intervention for diabetes on glycaemic control: a meta-analysis. Diabet Med. 2011 Apr;28(4):455-63. doi: 10.1111/j.1464-5491.2010.03180.x. PMID 21392066
- [Background] Mulvaney SA, Ritterband LM, Bosslet L. Mobile intervention design in diabetes: review and recommendations. Curr Diab Rep. 2011 Dec;11(6):486-93. doi: 10.1007/s11892-011-0230-y. PMID 21960031
- [Background] Wei J, Hollin I, Kachnowski S. A review of the use of mobile phone text messaging in clinical and healthy behaviour interventions. J Telemed Telecare. 2011;17(1):41-8. doi: 10.1258/jtt.2010.100322. Epub 2010 Nov 19. PMID 21097565
- [Background] Krishna S, Boren SA, Balas EA. Healthcare via cell phones: a systematic review. Telemed J E Health. 2009 Apr;15(3):231-40. doi: 10.1089/tmj.2008.0099. PMID 19382860
- [Background] Lee E, Tatara N, Arsand E, Hartvigsen G. Review of mobile terminal-based tools for diabetes diet management. Stud Health Technol Inform. 2011;169:23-7. PMID 21893707
- [Background] Quinn CC, Shardell MD, Terrin ML, Barr EA, Ballew SH, Gruber-Baldini AL. Cluster-randomized trial of a mobile phone personalized behavioral intervention for blood glucose control. Diabetes Care. 2011 Sep;34(9):1934-42. doi: 10.2337/dc11-0366. Epub 2011 Jul 25. PMID 21788632
- [Background] Whitehead L, Seaton P. The Effectiveness of Self-Management Mobile Phone and Tablet Apps in Long-term Condition Management: A Systematic Review. J Med Internet Res. 2016 May 16;18(5):e97. doi: 10.2196/jmir.4883. PMID 27185295
- [Background] Holmen H, Torbjornsen A, Wahl AK, Jenum AK, Smastuen MC, Arsand E, Ribu L. A Mobile Health Intervention for Self-Management and Lifestyle Change for Persons With Type 2 Diabetes, Part 2: One-Year Results From the Norwegian Randomized Controlled Trial RENEWING HEALTH. JMIR Mhealth Uhealth. 2014 Dec 11;2(4):e57. doi: 10.2196/mhealth.3882. PMID 25499872
- [Background] Waki K, Fujita H, Uchimura Y, Omae K, Aramaki E, Kato S, Lee H, Kobayashi H, Kadowaki T, Ohe K. DialBetics: A Novel Smartphone-based Self-management Support System for Type 2 Diabetes Patients. J Diabetes Sci Technol. 2014 Mar;8(2):209-215. doi: 10.1177/1932296814526495. Epub 2014 Mar 13. PMID 24876569
- [Background] Anarte Ortiz MT, Caballero FF, Ruiz de Adana MS, Rondan RM, Carreira M, Dominguez-Lopez M, Machado A, Gonzalo-Marin M, Tapia MJ, Valdes S, Gonzalez-Romero S, Soriguer FC. Development of a new fear of hypoglycemia scale: FH-15. Psychol Assess. 2011 Jun;23(2):398-405. doi: 10.1037/a0021927. PMID 21381839